CLINICAL TRIAL: NCT00144937
Title: A Randomized Controlled Trial Comparing Usual Care With a Multifactorial Intensified Intervention on Cardiovascular Risk Factors in Subjects With Arterial Peripheral Disease With and Without Diabetes. The Taulí Intervention Program (TIP).
Brief Title: Multifactorial Intervention on Cardiovascular Risk Factors in Subjects With Peripheral Arterial Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Sabadell (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 2003020
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Peripheral Arterial Disease; Hypercholesterolemia; Hypertension; Diabetes Mellitus; Smoking
MeSH Terms: conditions — Peripheral Arterial Disease; Hypercholesterolemia; Hypertension; Diabetes Mellitus; Smoking | interventions — Exercise

INTERVENTIONS:
Drug: Stepwise therapy for dyslipidemia, hypertension and diabetes
Behavioral: Dietary recommendations
Behavioral: Increase in physical activity
Behavioral: Smoking cessation

SUMMARY:
The purpose of this study was to evaluate whether an intensified multifactorial intervention program about cardiovascular risk factors in subjects with peripheral arterial disease (with and without diabetes mellitus), can improve the control of these factors (mainly hypercholesterolemia and hypertension) in relation to the habitual care

DETAILED DESCRIPTION:
Subjects with peripheral arterial disease show an increased cardiovascular risk. It is thought that improving control of cardiovascular risk factors (hypercholesterolemia, hypertension, diabetes, smoking) could be beneficial in reducing their cardiovascular risk. However, usual care of these subjects (mainly at primary care) is not associated with an optimal control of such cardiovascular risk factors. We hypothesise that an intensive multifactorial treatment in a Cardiovascular Risk Unit could improve control of these cardiovascular risk factors. To test this hypothesis we perform a controlled, randomized, open, parallel trial. Subjects are recruited at the Vascular Surgery Unit and are randomised into two groups: 1. usual care (control group); 2. intensive care (intervention group). Randomization is stratified for the presence/absence of diabetes mellitus and with the use of sealed envelopes. Patients assigned to receive usual care (general practitioner with the possibility of being referred to specialists) are compared to those assigned to undergo intensive multifactorial intervention. This intervention involves strict treatment goals (LDL-cholesterol < 100 mg/dl, blood pressure < 130/80, HbA1c < 7 %, no smoking) to be achieved through behavior modification (diet, physical activity, smoking cessation) and a stepwise introduction of pharmacologic therapy for hypercholesterolemia, hypertension and diabetes. This multifactorial intervention is overseen by a multidisciplinary team (endocrinologist, nurse, and dietitian) at the Hospital of Sabadell (Corporación Parc Taulí). The treatment goals are the same for the usual care group and general practitioners caring patients included in this study are informed of these strict treatment goals. Patients in the intensive-therapy receive 6 scheduled individual consultations in one year (baseline and 2,4, 6 and 9 months after their inclusion).Primary and secondary outcomes are evaluated at 12 months after their inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Arm-ankle index < 0.85 and > 0.40 in at least one leg

Exclusion Criteria:

* Advanced peripheral arterial disease (arm-ankle index < 0.40 or amputation)
* Peripheral arterial disease of non-atherosclerotic origin (e.g. vasculitis)
* Heart failure (NYHA III or IV)
* End-stage renal disease
* Atrial fibrillation
* Active peptic ulcer disease
* Blood coagulation disorders
* Platelets disorders
* Cancer
* History of rhabdomyolysis
* Treatment with immunosuppressant agents (e.g. cyclosporine, glucocorticoids)
* Excessive intake of alcohol (> 280 gr/week)
* Institutionalized patients

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Lowering of LDL cholesterol concentrations and blood pressure levels (at 12 months). Increase in use of antiplatelet agents (at 12 months)

SECONDARY OUTCOMES:
Decrease in basal glycaemia and HbA1c(only subjects with diabetes)
Lowering of serum triglycerides and total cholesterol.
Increase in serum HDL cholesterol
Improvement in cardiovascular risk (Framingham Score and UKPDS engine)
Weight reduction
Increase in physical activity
Changes in dietary intake
Smoking cessation
Improvement in health-related quality of life (SF-36)
Improvement of intermittent claudication
Improvement of arm-ankle index
Effect of control of cardiovascular risk factors on metabolic and inflammatory markers associated with cardiovascular disease
Changes in serum concentrations of hepatic enzymes
Changes in use of statins and fibrates
Changes in use of antihypertensive drugs and hypoglycemic agents
Cardiovascular events
All the above-mentioned primary and secondary outcomes will be evaluated at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: José-Miguel González-Clemente, MD, PhD, Principal Investigator — Department of Diabetes, Endocrinology and Nutrition. Hospital de Sabadell; Dídac Mauricio, MD, PhD, Study Chair — Department of Diabetes, Endocrinology and Metabolism. Hospital de Sabadell
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain